CLINICAL TRIAL: NCT03552445
Title: Immunogenicity and Safety of a Tetanus-diphtheria Vaccine and a 13-valent Pneumococcal Conjugate Vaccine After Concomitant Vaccination in ≥50-year-old Adults
Brief Title: Immunogenicity and Safety of a Tetanus-diphtheria Vaccine and a 13-valent Pneumococcal Conjugate Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Joon Young Song, Professor, Korea University Guro Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2013GR0005
Record Dates: First submitted 2018-05-17; First posted 2018-06-11 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-05

CONDITIONS: Tetanus; Diphtheria; Pneumococcal Infections
MeSH Terms: conditions — Tetanus; Diphtheria; Pneumococcal Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tetanus-diphtheria (Td) and PCV13 (Active Comparator)
  Interventions: Biological: Tetanus-diphtheria (Td) and PCV13
- PCV13 alone (Active Comparator)
  Interventions: Biological: PCV13 alone
- Td alone (Active Comparator)
  Interventions: Biological: Td alone

INTERVENTIONS:
Biological: Tetanus-diphtheria (Td) and PCV13 — 154 concomitant Td-PCV13 recipients: one dose of each vaccine administered on Day 0
  Arms: Tetanus-diphtheria (Td) and PCV13
Biological: PCV13 alone — 154 PCV13 recipients: one vaccine injection administered on Day 0
  Arms: PCV13 alone
Biological: Td alone — 437 Td recipients: one vaccine injection administered on Day 0
  Arms: Td alone

SUMMARY:
When two or more vaccines are administered concurrently, there is a concern on vaccine interaction, which can either enhance or suppress immune response to vaccine antigens. This study is designed to evaluate the immunogenicity and safety of tetanus-diphtheria (Td) and pneumococcal vaccines after concomitant administration in adults aged 50 years and older.

DETAILED DESCRIPTION:
Vaccination would be the most effective strategy to prevent diverse infectious diseases. Actually, The World Health Organization (WHO) estimate that vaccination averts 2-3 million deaths per year. In adults, several vaccines are recommended based on age and medical conditions if they have not receive vaccination before, and lack evidence of past infection: influenza, measles-mumps-rubella (MMR), varicella, human papilloma virus (HPV), tetanus-diphtheria (Td), pneumococcl vaccines and etc. In particular, when the patient visits a vaccination clinic, Td and the pneumococcal vaccines are commonly administered at the same time. In this study, we aimed to evaluate the immunogenicity and safety of Td vaccine and PCV13 after concomitant administration in adults aged 50 years. This single-center, open label randomized trial was conducted (Clinical Trial Number - NCT02215863) at Korea University Guro Hospital from November 2013 to April 2016. Adults ≥50 years of age were randomized in a 1:1:1 ratio to receive Td + PCV13 (Group 1), PCV13 alone (Group 2) or Td alone (Group 3).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥50 years who signed the informed consent

Exclusion Criteria:

* history of S. pneumoniae infection within the previous 5 years
* previous pneumococcal vaccination
* previous tetanus-diphtheria (Td) vaccination within the last 10 years
* known immunodeficiency or immunosuppressant use or coagulation disorders

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 462 (Actual)
Dates: Start 2013-11-01 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Tetanus antibody titers at day 28 post-vaccination | 4 weeks after vaccination
  IgG antibody titers by enzyme linked immunosorbent assay (ELISA) Seroprotection rate: percentage of subjects with a post-vaccination antibody levels ≥0.1 IU/mL
Diphtheria antibody titers at day 28 post-vaccination | 4 weeks after vaccination
  IgG antibody titers by enzyme linked immunosorbent assay (ELISA)
Tetanus seroprotection rate at day 28 post-vaccination | 4 weeks after vaccination
  Proportion of IgG antibody titers ≥0.1 IU/mL
Diphtheria seroprotection rate at day 28 post-vaccination | 4 weeks after vaccination
  Proportion of IgG antibody titers ≥0.1 IU/mL

SECONDARY OUTCOMES:
Opsonophagocytic assay (OPA) titers for PCV13 | 4 weeks after vaccination
  Four capsule serotypes: 1, 5, 18C and 19A

OTHER OUTCOMES:
Frequency and duration of local and systemic adverse events | During 4 weeks after vaccination
  The safety profiles of co-administration of Td and PCV13 will be compared to those of single vaccination.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Song JY, Cheong HJ, Noh JY, Choi MJ, Yoon JG, Lee SN, Kang SH, Jeong EJ, Jo YM, Kim WJ. Immunogenicity and safety of a tetanus-diphtheria vaccine and a 13-valent pneumococcal conjugate vaccine after concomitant vaccination in >/= 50-year-old adults. BMC Infect Dis. 2018 Dec 5;18(1):628. doi: 10.1186/s12879-018-3479-9. PMID 30518331